CLINICAL TRIAL: NCT04540276
Title: Intraoperative Hyperoxia and MINS: A Post Hoc Analysis From the VISION Study Database
Brief Title: Intraoperative Hyperoxia and MINS
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University Hospital Bispebjerg and Frederiksberg (Other)
Collaborators: Population Health Research Institute (Other)
Responsible Party: Principal Investigator, Sofie Pedersen, MD, PhD-student at Dept. of Anesthesia and Intensive Care, University Hospital Bispebjerg and Frederiksberg
Other Study IDs: Hyperoxia and MINS
Record Dates: First submitted 2020-08-31; First posted 2020-09-07 (Actual); Last update posted 2021-02-04 (Actual); Status verified 2021-02

CONDITIONS: Hyperoxia; Myocardial Infarction; Myocardial Injury
MeSH Terms: conditions — Hyperoxia; Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Inspiratory oxygen fraction — Median inspiratory oxygen fraction during general anesthesia

SUMMARY:
Oxygen therapy is administered to all patients during general anesthesia to maintain tissue oxygenation and prevent hypoxia and ischemia. However, liberal use of oxygen may lead to hyperoxia and some studies suggest that supranormal levels of arterial oxygen saturation may lead to complications. In this post hoc substudy of the VISION cohort, we plan to assess the association between perioperative inspired oxygen fraction (FiO2) and myocardial injury after non-cardiac surgery (MINS).

DETAILED DESCRIPTION:
Patients will be divided into five groups of median intraoperative FiO2 (quintiles), in which baseline characteristics and outcomes will be illustrated.

The odds ratio (OR) for the primary and secondary outcomes will be calculated in a logistic regression analysis with median FiO2 (continuous variable) as independent variable.

Analyses are performed with multiple logistic regression with adjustment for the following potentially confounding variables:

Age ≥75 years. Male sex. Current atrial fibrillation. History of diabetes. History of congestive heart failure. History of coronary artery disease. History of recent (i.e., < 6 months) high-risk coronary artery disease. History of stroke. History of peripheral vascular disease. History of hypertension. Preoperative eGFR (<30 vs. 30-44 vs. 45-59 vs. ≥60 mL/min/1.73m2). Low-risk surgery. Duration of surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients entered in the VISION database, aged 18 years or above, undergoing noncardiac surgery in general anesthesia.

Exclusion Criteria:

* Patients with unobtainable data on perioperative FiO2.
* Patients with unobtainable data on postoperative troponin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients entered in the VISION database, undergoing noncardiac surgery in general anesthesia.
Sampling Method: Probability Sample
Enrollment: 7700 (Estimated)
Dates: Start 2018-02-04 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2021-03-01 (Estimated)

PRIMARY OUTCOMES:
Myocardial injury after non-cardiac surgery (MINS) | Within 30 days after surgery.
  Number of participants with MINS in the specified oxygen groups. MINS is defined as either ischemic troponin elevation or myocardial infarction after non-cardiac surgery.

SECONDARY OUTCOMES:
All-cause mortality | Within 30 days after surgery
  Number of deaths within 30 days after surgery
Myocardial infarction | Within 30 days after surgery
  Number of participants with myocardial infarction within 30 days after surgery
MINS | Within 30 days after surgery
  Number of participants with MINS not fulfilling the fourth universal definition of myocardial infarction
Rehospitalization for vascular reasons | Within 30 days after surgery
  Number of participants rehospitalized for vascular reasons within 30 days after surgery
Pneumonia | Within 30 days after surgery
  Number of participants with pneumonia within 30 days after surgery

OTHER OUTCOMES:
Vascular mortality | Within 30 days after surgery
  Number of vascular deaths within 30 days after surgery
Non-fatal cardiac arrest | Within 30 days after surgery
  Number of participants with non-fatal cardiac arrest within 30 days after surgery
Cardiac revascularization procedure | Within 30 days after surgery
  Number of participants undergoing cardiac revascularization procedure within 30 days after surgery
Pulmonary embolism | Within 30 days after surgery
  Number of participants with pulmonary embolism within 30 days after surgery
New-onset clinically important atrial fibrillation | Within 30 days after surgery
  Number of participants with new-onset clinically important atrial fibrillation within 30 days after surgery
Peripheral arterial thrombosis | Within 30 days after surgery
  Number of participants with peripheral arterial thrombosis within 30 days after surgery
Severe sepsis or septic shock | Within 30 days after surgery
  Number of participants with severe sepsis or septic shock within 30 days after surgery
Surgical wound infection | Within 30 days after surgery
  Number of participants with surgical wound infection defined as surgical incision infection or surgical abscess
Deep venous thrombosis | Within 30 days after surgery
  Number of participants with deep venous thrombosis within 30 days after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Christian S. Meyhoff, MD, PhD, Principal Investigator — University hospital Bispebjerg Frederiksberg; PJ Devereaux, MD, PhD, Study Chair — Population Healt Research Institute
Locations (8):
- Cleveland Clinic, Cleveland, Ohio, United States
- Walter C. Mackenzie Health Sciences Centre, Edmonton, Canada
- Prince of Wales Hospital, Hong Kong, China
- Foundation CardioInfanil, Bogotá, Colombia
- Bispebjerg Hospital, Copenhagen, NV, Denmark
- Christian Medical College, Ludhiāna, India
- University Malaya Medical Centre, Kuala Lumpur, Malaysia
- Inkosi Albert Luthuli Hospital, Durban, South Africa